CLINICAL TRIAL: NCT03056118
Title: Optimal Duration of Clopidogrel After Implantation of Second-Generation Drug-Eluting Stents (OPTIMA-C)
Brief Title: Optimal Duration of Clopidogrel in Second-Generation Drug-Eluting Stents
Acronym: OPTIMA-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Hyuck moon Kwon, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 3-2011-0054
Record Dates: First submitted 2017-02-08; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Ischemic Heart Disease
Keywords: OPTIMA-C
MeSH Terms: conditions — Myocardial Ischemia | interventions — Dual Anti-Platelet Therapy; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 6-month dual anti-platelet therapy (Experimental): maintain dual anti-platelet agents for 6 months
  Interventions: Drug: 6-month dual anti-platelet therapy
- 12-month dual anti-platelet therapy (Active Comparator): maintain dual anti-platelet agents for 12 months
  Interventions: Drug: 12-month dual anti-platelet therapy
- Zotarolimus eluting stent arm (Active Comparator): implant with zotarolimus eluting stent (Resolute Integrity)
  Interventions: Device: Zotarolimus eluting stent
- Biolimus eluting stent arm (Active Comparator): implant with biolimus eluting stent (Biomatrix)
  Interventions: Device: Biolimus eluting stent

INTERVENTIONS:
Drug: 6-month dual anti-platelet therapy — Aspirin and P2Y12 inhibitor after percutaneous coronary intervention continues for 6 months
  Other Names: Aspirin and Clopidogrel
  Arms: 6-month dual anti-platelet therapy
Drug: 12-month dual anti-platelet therapy — Aspirin and P2Y12 inhibitor after percutaneous coronary intervention continues for 12 months
  Other Names: Aspirin and Clopidogrel
  Arms: 12-month dual anti-platelet therapy
Device: Zotarolimus eluting stent — Zotarolimus eluting stent is applied to coronary stenotic lesion
  Arms: Zotarolimus eluting stent arm
Device: Biolimus eluting stent — Biolimus eluting stent is applied to coronary stenotic lesion
  Arms: Biolimus eluting stent arm

SUMMARY:
Investigators try to assess the safety of 6-months or 12-months maintenance of dual antiplatelet therapy (DAPT, aspirin + clopidogrel) in patients undergoing percutaneous coronary intervention using the Zotarolimus-eluting, Resolute Integrity™ stent (Medtronic Vascular Inc, Santa Rosa, CA) or the BioMatrix™ stent (Biosensors. Singapore).

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) has proven the most effective treatment in reducing thrombotic complications after drug eluting stent (DES) implantation. Although the optimal duration of antiplatelet therapy is still under investigation, late stent thrombosis (ST) with DES has pushed the recommendation for duration of clopidogrel therapy for one year or more, in patients without risks for bleeding. However, recent controversies regarding the risk of stent thrombosis in patients receiving DES has brought up the issue of the appropriate duration of antiplatelet therapy after percutaneous coronary intervention, and a recent study reported that the use of extended DAPT for a period longer than 12 months in patients who had received DES was not significantly more effective than aspirin monotherapy in reducing the rate of myocardial infarction (MI) or death for cardiac causes.

Zotarolimus-eluting stent (Resolute Integrity™) and biolimus-eluting stent with biodegradable polymer system (BioMatrix™) share several similarities. Both stents are flexible thin strut stents eluting sirolimus-analogue drugs targeting at mammalian target of rapamycin. The advantages that Resolute Integrity™ stent strut is quite thin and coated with highly biocompatible polymer and BioMatrix™ stent has the abluminal drug coating system with biodegradable polymer might provide clinical studies showing that both stents are quite safe as well as efficacious. Moreover, recent report showed that continuation of clopidogrel for only 3 months after implantation of Endeavor stent seems to be safe in low-to-moderate coronary artery risk group. Based on these clinical evidences, the duration of DAPT continuation for 12 months or less after implantation of Resolute Integrity™ or BioMatrix™ stent, 'the second generation DES', would be safe, however, there are no data available about this. Therefore, the purpose of this study is to assess the safety of 6-months or 12-months maintenance of DAPT in patients undergoing percutaneous coronary intervention (PCI) using Resolute Integrity™ or BioMatrix™ stent.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 20 years of age.
2. Subject must have evidence of myocardial ischemia (e.g. stable angina, non-ST elevation acute coronary syndrome, silent ischemia, positive functional study or a reversible changes in the electrocardiogram (ECG) consistent with ischemia).
3. Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving the Resolute Integrity or BioMatrix stent and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

Exclusion Criteria:

1. Acute ST elevation myocardial infarction
2. The patient has a known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, zotarolimus, biolimus, contrast media
3. Clinical conditions requiring systemic immune suppression over 2 weeks or anti-cancer therapy
4. Prior history of the following presentations: Thromboembolic disease, Stent thrombosis
5. Pregnant women or women with childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
6. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions.
7. Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
8. Current known current platelet count < 100,000 cells/mm3 or Hgb <10 g/dL.
9. Non-cardiac co-morbid conditions are present with life expectancy < 1 year or that may result in protocol non-compliance (per site investigator's medical judgment
10. Patients with left ventricular ejection fraction < 35%
11. Patients with cardiogenic shock
12. Creatinine level > 2.4mg/dL
13. Severe hepatic dysfunction (aspartate aminotransferase and/or alanine aminotransferase ≥ 3 times upper normal reference values)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1368 (Actual)
Dates: Start 2011-05-02 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-09-07 (Actual)

PRIMARY OUTCOMES:
A composite of major adverse cardiac events (MACE; cardiac death, target vessel MI and ischemia driven-target lesion revascularization; TLR) | 12 months
  1. Cardiac death: Any death due to proximate cardiac cause (eg, MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death.
  2. MI Classification and Criteria for Diagnosis is defined by the Academic Research Consortium
  3. TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLRs should be classified prospectively as clinically indicated* or not clinically indicated by the investigator prior to repeat angiography. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Hyuck moon Kwon, Principal Investigator — Gangnam Severance Hospital

IPD SHARING:
Plan to Share IPD: Yes
If PI and scientific committee approve to share individual participant data to other researchers.

REFERENCES:
- [Derived] Jang JY, Jung HW, Lee BK, Shin DH, Kim JS, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Park KW, Gwon HC, Kim HS, Kwon HM, Jang Y. Impact of PRECISE-DAPT and DAPT Scores on Dual Antiplatelet Therapy Duration After 2nd Generation Drug-Eluting Stent Implantation. Cardiovasc Drugs Ther. 2021 Apr;35(2):343-352. doi: 10.1007/s10557-020-07008-7. PMID 32588238